CLINICAL TRIAL: NCT06355635
Title: Evaluation of Application and Monitoring of Vasoactive and Inotrope Drugs in Non-cardiac Surgery Patients
Brief Title: Application and Monitoring of Vasoactive and Inotrope Drugs
Acronym: Vasin
Status: Recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: JohannesGUVA
Record Dates: First submitted 2023-06-16; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Hemodynamic Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Choice and Monitoring — current practive of vasoactive and inotrope drugs
  Other Names: current practice

SUMMARY:
The investigators aimed to establish current practice of application and monitoring of vasoactive and inotrope Drugs in non-cardiac surgery patients.

DETAILED DESCRIPTION:
This survey provides a current update on a variety of cardioactive and vasoactive drugs at non-cardiac surgery patients in germany.

ELIGIBILITY:
Inclusion Criteria:

* all anesthesiologists of germany

Exclusion Criteria:

* not completely responses

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All Anesthesiologists
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
current practice of correct application and monitoring of vasoactive and inotrope Drugs | through study completion, an average of 2 months
  physiological parameter, Units on a scale

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, Principal Investigator — University Medical Centre
Locations (1):
- Department of Anaesthesiology;, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No